CLINICAL TRIAL: NCT02997891
Title: Change of Cognitive Performance for Older People Through Artificial Hip Replacement Implantation [German Title: Veränderungen Der Kognitiven Leistungsfähigkeit älterer Menschen Durch Hüft-TEP Implantation]
Brief Title: Change of Cognitive Performance Through Hip Replacement
Acronym: KogniTEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Stiftung Endoprothetik (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKE 0545/110
Record Dates: First submitted 2016-07-14; First posted 2016-12-20 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis, Hip
Keywords: cognition; hip replacement; physical activity; quality of life; psychological distress
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intervention group: Patients with primary, unilateral hip osteoarthritis in inpatient orthopedic acute treatment, who have a medical indication of a necessary artificial hip replacement implantation.
  Interventions: Diagnostic Test: everyday activity; Diagnostic Test: cognitive performance
- control group: Volunteers without chronic pain. As a control condition for comparing the variation in cognitive performance and everyday activity the investigators use a group of pain-free and mobility-unrestricted subjects, who do not receive or have an artificial hip.
  Interventions: Diagnostic Test: everyday activity; Diagnostic Test: cognitive performance

INTERVENTIONS:
Diagnostic Test: everyday activity — To objectively quantify the everyday activity, there are a variety of instruments, without a currently gold standard. Therefore, in addition the investigators use objectified measurement parameters with the aid of a pedometer (GARMIN vivofit) on every three measuring time points (before surgery, 3 months after surgery, 6 months after surgery).
Diagnostic Test: cognitive performance — Standardized neuropsychological assessment methods are used to assess the cognitive performance. To assess the degree of mobility, health status and the physical activity standardized questionnaires are used.

SUMMARY:
The purpose of this study is to investigate the effectiveness of a hip arthroplasty for chronic pain, caused by a unilateral primary Coxartrhrose, regarding the cognitive performance. It is based on the hypothesis that the combination of chronic pain along with relative immobilization causes impairment of cognitive performance. The total hip replacement reduces pain, increases the mobility level and finally improves the cognitive performance.

DETAILED DESCRIPTION:
Studies have shown that cognitive performance, especially in the elderly is limited due to chronic pain. In a recent study, significantly less brain activity in various regions of the brain (the anterior cingulate cortex (ACC), insula and operculum, dorsolateral prefrontal cortex and orbitofrontal cortex) was detected in patients with unilateral primary coxarthrosis compared to a healthy control group. After eliminating the pain by the implantation of a total hip replacement, a significant increase in brain activity in the affected areas was observed in these patients. Whether this observation is accompanied by an effect on cognition, is not known and will be investigated in the proposed study. The purpose of this study is to investigate the effectiveness of a hip arthroplasty for chronic pain, caused by a unilateral primary Coxartrhrose, regarding the cognitive performance. It is based on the hypothesis that the combination of chronic pain along with relative immobilization causes impairment of cognitive performance. The total hip replacement reduces pain, increases the mobility level and finally improves the cognitive performance.

The main issue concerns the short and mid-term influence of hip replacement on cognitive performance in the perioperative care continuum in comparison to a control group that does not have chronic pain. To objectively quantify the everyday activity, there are a variety of instruments, without a currently gold standard. Therefore, in addition the investigators use objectified measurement parameters with the aid of a pedometer (GARMIN vivofit) on every three measuring time points (before surgery, 3 months after surgery, 6 months after surgery).

Standardized neuropsychological assessment methods are used to assess the cognitive performance. To assess the degree of mobility, health status and the physical activity standardized questionnaires are used.

Primary hypothesis: After implantation of an artificial hip replacement and reduction of experienced pain patients with primary coxarthrosis indicate an improvement of cognitive performance 3 and 6 month after surgery compared to the pre-surgical status. In addition, the investigators measure how severe the cognitive performance is reduced compared to a healthy control group prior to surgery and to what extend the cognitive performance is reversible in the aftermath.

ELIGIBILITY:
Inclusion Criteria:

* primary, unilateral coxarthrosis
* planning for hip replacement surgery in Bad Bramstedt

Exclusion Criteria:

* dementia / cognitive impairment (Mini Mental Status Test <25)
* chronic pain otherwise genesis
* reduced physical activity otherwise genesis
* lack of German language skills
* uncorrected serious impairment of vision or hearing
* serious additional psychiatric diagnoses (e.g. substance abuse / addiction)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients are enrolled in this study, who are diagnosed in the orthopedic clinic of Klinikum Bad Bramstedt or in the orthopedic clinic at University Medical Center Hamburg-Eppendorf. Study participants with the diagnosis of primary, unilateral coxarthrosis (ICD-10-GM: M16.1) are added consecutively in the intervention group, if they need a hip replacement because of their condition and decide to undergo this hip replacement in the orthopedic clinic of Klinikum Bad Bramstedt.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
attention and concentration performance (assessed by d2 Test of Attention) | Change from Baseline attention and concentration performance at 6 months
conceptual tracking, planning and flexibility (assessed by Trail Making Tests (Parts A and B) | Change from Baseline conceptual tracking, planning and flexibility at 6 months
semantic memory (assessed by FAS-Test [Verbal Fluency]) | Change from Baseline semantic memory at 6 months
verbal episodic memory (Rivermead Behavioural Memory Test (RBMT) - story recall subtest) subtest | Change from Baseline verbal episodic memory at 6 months
visuospatial constructional ability and visual memory (assessed by Rey-Osterrieth Complex Figure Test) | Change from Baseline visuospatial constructional ability and visual memory at 6 months

SECONDARY OUTCOMES:
subjective physical activity (assessed by Physical Activity Scale for the Elderly (PASE)) | Change from Baseline subjective physical activity at 6 months
objective physical activity (assessed by pedometer GARAMIN vivofit) | Change from Baseline objective physical activity at 6 months
anxiety (assessed by the Generalized Anxiety Disorder 7-Scale (GAD-7)) | Change from Baseline anxiety at 6 months
depression (assessed by the Patient Health Questionnaire (PHQ-9)) | Change from Baseline depression at 6 months
quality of life (assessed by the SF-12 health survey) | Change from Baseline quality of life at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Niemeier, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (2):
- Germany (2):
  - Klinikum Bad Bramstedt, Bad Bramstedt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Raecke R, Niemeier A, Ihle K, Ruether W, May A. Brain gray matter decrease in chronic pain is the consequence and not the cause of pain. J Neurosci. 2009 Nov 4;29(44):13746-50. doi: 10.1523/JNEUROSCI.3687-09.2009. PMID 19889986
- [Background] Rodriguez-Raecke R, Niemeier A, Ihle K, Ruether W, May A. Structural brain changes in chronic pain reflect probably neither damage nor atrophy. PLoS One. 2013;8(2):e54475. doi: 10.1371/journal.pone.0054475. Epub 2013 Feb 6. PMID 23405082